CLINICAL TRIAL: NCT06316011
Title: Magnetocardiography in the Identification and Risk Stratification of Patients With Acute Chest Pian
Brief Title: MCG for Risk Stratifications of Patients With Chest Pain
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Chongqing Emergency Medical Center (Other); Weifang People's Hospital (Other); Linyi People's Hospital (Other); Weihai Central Hospital (Other); Jining First People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First People's Hospital of Hangzhou (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Qianfoshan Hospital (Other); Heze Municipal Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: MCG-chestpain
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Magnetocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training and testing cohort
  Interventions: Device: Magnetocardiography
- External validation cohort
  Interventions: Device: Magnetocardiography

INTERVENTIONS:
Device: Magnetocardiography — Magnetocardiography

SUMMARY:
This prospective cohort study is aimed at identification and risk stratification of patients who have symptoms of acute chest pain suspected with acute coronary syndrome （ACS） using Magnetocardiography （MCG）.

ELIGIBILITY:
Inclusion Criteria:

* Those with suspected ACS who presented with symptoms of acute chest pain.
* Signed informed consent.

Exclusion Criteria:

* Those with known structural heart disease such as cardiomyopathy and valvular disease;
* Those with atrial fibrillation, supraventricular tachycardia, atrioventricular block and other arrhythmias that have not returned to normal;
* Those who have chest pain with known pulmonary embolism or aortic coarctation;
* Those who are thought to be incapable of completing the MCG examination by an attending physician (or physician with higher qualifications) due to unstable clinical conditions, metal implants, etc;
* Those who are unable to perform magnetocardiography examinations due to claustrophobia, etc., or those who fail to receive magnetocardiography examination;
* Those with malignant tumors;
* Pregnant or lactating women.
* Those with acute or critical illnesses of other systems, such as acute or severe respiratory illnesses, marked abnormalities in liver function or kidney function.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient who suffers from cardiogenic chest pain suspected with acute coronary syndrome （ACS）.
Sampling Method: Non-Probability Sample
Enrollment: 3620 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of MCG for the detection and risk stratification in high-risk patients with chest pain | from the date of enrollment until the date of discharge, up to 30 days
  Establishing an algorithm model of MCG in identifying high-risk cardiogenic chest pain, the efficacy of the model was assessed by sensitivity, specificity, accuracy, positive predictive value, negative predictive value, and AUC, etc.
Efficacy of MCG for the detection and risk stratification in low-risk patients with chest pain | from the date of enrollment until the date of discharge, up to 30 days
  Establishing an algorithm model of MCG in identifying low-risk cardiogenic chest pain, the efficacy of the model was assessed by sensitivity, specificity, accuracy, positive predictive value, negative predictive value, and AUC, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Professor, Principal Investigator — Qliu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China